CLINICAL TRIAL: NCT00700388
Title: Multicenter Controlled Trial on Efficacy of TPEP Device in Adult Patients With Chronic Hypersecretion
Brief Title: Efficacy of Temporary Positive Expiratory Pressure (TPEP) in Chronic Hypersecretion
Acronym: UNIKO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Villa Pineta Hospital (Other)
Collaborators: University of Modena and Reggio Emilia (Other)
Responsible Party: Prof. Enrico Clini, University of Modena - Villa Pineta Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 69/08
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2010-01

CONDITIONS: Chronic Hypersecretions
Keywords: Chronic bronchitis; COPD; Bronchiectasis
MeSH Terms: conditions — Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive; Bronchiectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): TPEP added to conventional manually assisted breathing techniques (MABT)
  Interventions: Device: TPEP device (UNIKO)
- 2 (Active Comparator): Manually assisted breathing techniques (MABT) alone
  Interventions: Procedure: MABT (Manually assisted breathing techniques)

INTERVENTIONS:
Device: TPEP device (UNIKO) — This technique is mainly based on a continuous low-pressure insufflation in the airways, which is likely to reduce (or even avoid) the potential pressure-related damages of other commonly used devices. This device should be used only in those individuals who are showing a normal competence of their cough reflex, thus it should be considered as a means which may help those techniques normally adopted for the individual's bronchial hygiene.
  Other Names: UNIKO
  Arms: 1
Procedure: MABT (Manually assisted breathing techniques) — Conventionally manually assisted breathing techniques
  Other Names: MABT
  Arms: 2

SUMMARY:
Mechanical devices to increase the individual's bronchial hygiene are commonly used in patients with chronic retention of secretions and abnormal cough reflex. In this clinical context a new technology (namely TPEP® - Temporary Positive Expiratory Pressure) has been recently developed with the aim to improve the respiratory condition in patients suffering from chronic respiratory diseases. This trial has the aim to assess the clinical efficacy of TPEP in patients with chronic hypersecretion and airways obstruction, but with a normal competence of the cough reflex

DETAILED DESCRIPTION:
This is a single-blind multicentre controlled randomized trial with consecutive recruitment. Randomization list by blocks will be available. Group comparison will be made between active therapies including TPEP added to conventional MABT (Intervention) or MABT alone (Control). Active therapy will last 10 consecutive daily sessions in both groups.

Primary outcome

Efficacy comparison on change in:

a.arterial oxygenation (as assessed by PaO2/FiO2 ratio and/or SatO2 index)

Secondary outcomes

Efficacy comparison on change in:

1. Sputum characteristics
2. Daily sputum volume
3. Perceived sensation
4. Lung functions (as assessed by spirometry and RM strength)

ELIGIBILITY:
Inclusion Criteria:

* chronic hypersecretion as defined by > 30 mL/die sputum production (7)
* chronic airway obstruction (by definition)
* COPD, bronchiectasis, asthma, cystic disease, etc. with or without chronic respiratory failure
* adulthood
* smoking or non-smoking habit
* Peak Cough Expiratory Flow > 150 L*min-1 (5)
* willingness to participate

Exclusion Criteria:

* childhood
* presence of acute exacerbation
* severe concomitant cardiovascular diseases
* concomitant neoplastic diseases
* non compliance/adherence to TPEP
* concomitant use of chronic mechanical ventilation
* use of amynophyllines and/or any active drugs (e.g. N-Acetyl-Cysteine)

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
arterial oxygenation (as assessed by PaO2/FiO2 ratio and/or SatO2 index) | Day 10

SECONDARY OUTCOMES:
Sputum volume | Day 1 to 10
Sputum characteristics | Day 1 to 10
Individual's perceived sensation (VAS scale) | Day 1 to 10
Lung function (volumes and respiratory muscle performance) | Day 1 - 3 - 10

CONTACTS AND LOCATIONS:
Overall Officials: Enrico M. Clini, MD, Study Director — University of Modena - Villa Pineta Hospital; Nicolino Ambrosino, MD, Study Chair — AOU Pisana - Cisanello (Pisa)
Locations (6):
- Italy (6):
  - Fondazione Maugeri IRCCS, Lumezzane, Brescia
  - Villa Pineta Hospital, Pavullo nel Frignano, Modena
  - Fondazione Maugeri IRCCS, Veruno, Novara
  - Centro Riabilitazione Auxilium Vitae, Volterra, Pisa
  - Ospedale San Raffaele IRCCS, Volterra, Roma
  - Ospedale San Giuseppe - Riabilitazione Specialistica, Milan